CLINICAL TRIAL: NCT00927420
Title: Epidemiological Study to Evaluate Adherence to Treatment in Bipolar Disorder: Adherence Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NES-DUM-2009/1
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; adherence; treatment; real life practice
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed with bipolar disorder I or II (DSM-IV) in ambulatory settings

SUMMARY:
The purpose of this study is to estimate adherence to treatment in bipolar patients, to characterize patients based on adherence degree and to describe the variables linked to poor adherence to treatment in real-life practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bipolar disorder I or II DSM-IV
* Patients treated with at least one oral antipsychotic
* Subjects able to read and write

Exclusion Criteria:

* Patients participating in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bipolar disorder I or II (DSM-IV) in ambulatory settings
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Morisky-Green Scale | Once, at the visit moment
Drug Attitude Inventory Scale (DAI-10) | Once, at the visit moment

SECONDARY OUTCOMES:
Clinical Global Impressions for Bipolar illness-modified (CGI-BP-M) | Once, at the visit moment
Functioning Assessment Short Test (FAST) | Once, at the visit moment

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Gil, Study Director — AstraZeneca Spain EpidemiologyValue Demonstration Unit
Locations (24):
- Spain (24):
  - Research Site, Las Palmas, Gran Canarias
  - Research Site, Calahorra, La Rioja
  - Research Site, Langreo, Principality of Asturias
  - Research Site, San Cristóbal de La Laguna, Tenerife
  - Research Site, Alicante
  - Research Site, Almería
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Elche
  - Research Site, León
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Ourense
  - Research Site, Palma de Mallorca
  - Research Site, Salamanca
  - Research Site, Seville
  - Research Site, Toledo
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Vitoria-Gasteiz
  - Research Site, Zaragoza